CLINICAL TRIAL: NCT01677949
Title: A Phase II Trial Investigating Clofarabine, Cyclophosphamide and Etoposide for Minimal Residual Disease Positive Acute Leukemia
Brief Title: Clofarabine, Cyclophosphamide and Etoposide for Minimal Residual Disease Positive Acute Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011LS158; HM2012-05 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2012-08-28; First posted 2012-09-03 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2016-04

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Clofarabine; Etoposide; etoposide phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALL patients receiving transplant (Experimental): Patients intent on receiving an allogeneic hematopoietic cell transplantation (allo-HCT) with the diagnosis of acute lymphoblastic leukemia (ALL) along with Clofarabine, Etoposide and Cyclophosphamide.
  Interventions: Drug: Clofarabine; Drug: Etoposide; Drug: Cyclophosphamide; Biological: allogeneic hematopoietic cell transplantation
- AML patients receiving transplant (Experimental): Patients intent on receiving an allogeneic hematopoietic cell transplantation (allo-HCT) with the diagnosis of acute myeloid leukemia (AML) along with Clofarabine, Etoposide and Cyclophosphamide.
  Interventions: Drug: Clofarabine; Drug: Etoposide; Drug: Cyclophosphamide; Biological: allogeneic hematopoietic cell transplantation

INTERVENTIONS:
Drug: Clofarabine — Days 1-5: Clofarabine 30 mg/m^2 for 0-30 years of age or 20 mg/m^2 for > 30 years of age intravenously (IV) over 2 hours
  Other Names: Clolar
Drug: Etoposide — Days 1-5: Etoposide 100mg/m^2 IV over 2 hours
  Other Names: Eposin; Etopophos; Vepesid; VP-16
Drug: Cyclophosphamide — Days 1-5: Cyclophosphamide 300 mg/m^2 as a 30-60 minute infusion
  Other Names: Cytoxan
Biological: allogeneic hematopoietic cell transplantation — Between Days 28 and 42: infused independent of this study
  Other Names: allo-HCT

SUMMARY:
Study Design:

This is a two-stage Phase II trial investigating the efficacy of Clofarabine, Cyclophosphamide and Etoposide in acute leukemia patients with detectable minimal residual disease (MRD) prior to allo-HCT. The primary objective is to determine the impact of the study treatment in eliminating the presence of minimal residual disease without causing a significant delay of allo-HCT due to treatment related toxicity. The intent of this study is to allow patients to proceed to transplant (independent of this study) within 42 days of Day 1 of Clofarabine based therapy.

DETAILED DESCRIPTION:
Patients will be stratified at the time of enrollment based on diagnosis (ALL versus AML). Based on this two-stage optimal design, a maximum of 49 patients with ALL and a maximum of 49 patients with AML will be needed. For each disease cohort, 21 patients will be enrolled in stage 1. If at the end of stage 1, the criteria is met for activating stage 2 (based on success of clearing MRD, proceeding to transplant within 42 days and without excessive toxicity) for one or both groups, stage 2 will be activated with an additional 28 patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute lymphoblastic leukemia (ALL) or acute myeloid leukemia (AML) with <5% blasts in the bone marrow (M1) by morphology and that meets one of the following criteria:

  * Flow cytometric evidence of MRD (≥ 0.1% leukemic blasts for ALL or <5% leukemic blasts for AML detected in the bone marrow) OR
  * Molecular/cytogenetic evidence of disease (FISH or PCR methodology) performed within 7 days
  * AND with the intent of going on to an allogeneic hematopoietic cell transplantation (allo-HCT) independent of this study
* Age 0 to 60 years
* Karnofsky Performance Status ≥ 50% for patients 16 years and older and Lansky Play Score ≥ 50 for patients under 16 years of age
* Patients must have a life expectancy ≥ 8 weeks as determined by the enrolling investigator
* Have acceptable organ function as defined within 7 days of study registration:

  * Renal: creatinine clearance ≥70mL/min/1.73m2 or serum creatinine based on age/gender
  * Hepatic: aspartate aminotransferase (ALT) < 5 x upper limit of normal (ULN) and total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age
  * Cardiac: left ventricular ejection fraction ≥ 40% by echocardiogram (ECHO/MUGA)
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. At least 14 days must have elapsed from prior chemotherapy; at least 7 days must have elapsed since receiving biological therapy.

Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor and at least 14 days since pegfilgrastim (Neulasta®) administration.

* Sexually active females of child bearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment and for 2 months after the last dose of chemotherapy. Sexually active men must agree to use barrier contraceptive for the duration of treatment and for 2 months after the last dose of chemotherapy.
* Voluntary written consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care

Exclusion Criteria:

* Acute Promyelocytic Leukemia (APL)
* Active central nervous system (CNS) leukemia or known chloromatous disease
* Receiving or plans to receive concomitant chemotherapy, radiation therapy; immunotherapy or other anti-cancer therapy other than is specified in the protocol
* Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Pregnant or lactating. The agents used in this study are known to be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy.
* Known allergy to any of the agents or their ingredients used in this study

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of Patients Unable to Proceed to Transplantation | Between Day 30 and Day 42
  The primary endpoint of this study will be to determine the impact of Clofarabine, Cyclophosphamide and Etoposide on the conversion to an minimal residual disease (MRD) negative state at day 30 (<0.01% leukemic blasts by flow cytometry) or day 42 if day 30 marrow is un-evaluable due to hypocellularity per RECIST criteria as well as the ability of patients to reach allo-HCT without significant delay due to study treatment related toxicity. Unable to proceed to transplant by Day 42 will be considered unacceptable.

SECONDARY OUTCOMES:
Rate of Pre-Transplant Chemotherapy-Induced Aplasia | After Day 42
  defined as greater than 42 days after infusion of chemotherapy
Rate of Infectious Complications | Day 1 Through Day 30
Treatment-Related Mortality After Transplant | Day 100
  In the field of transplantation, toxicity is high and all deaths without previous relapse or progression are usually considered as related to transplantation.
Disease-Free Survival After Transplant | 1 Year
  The length of time after treatment ends that a patient survives without any signs or symptoms of that cancer or any other type of cancer. In a clinical trial, measuring the disease-free survival is one way to see how well a new treatment works.
Rate of Leukemic Relapse After Transplant | Day 100
  The return of disease after its apparent recovery/cessation.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Burke, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States